CLINICAL TRIAL: NCT04725812
Title: Complement Regulation to Undo Systemic Harm in Preeclampsia: The CRUSH Study
Brief Title: Complement Regulation to Undo Systemic Harm in Preeclampsia
Acronym: CRUSH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI moved institutions
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, S Ananth Karumanchi, Professor of Medicine, Cedars-Sinai Medical Center, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000039
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Preeclampsia; Severe Preeclampsia; Eculizumab; HELLP; HELLP Syndrome; HELLP Syndrome Second Trimester; Pregnancy Related; AHUS; PNH; Complement Regulatory Factor Defect; Complement Abnormality; HELLP Syndrome Third Trimester
MeSH Terms: conditions — Pre-Eclampsia; HELLP Syndrome | interventions — eculizumab

STUDY DESIGN:
Intervention Model Description: Single arm open label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eculizumab (Experimental): Twelve subjects in the interventional arm will receive eculizumab at an induction dose of 900mg IV weekly (q7 days) for 4 weeks followed by a dose of 1200mg IV at week 5. Thereafter, patients will receive a maintenance dose of 1200mg IV every two weeks (q14 days). The last dose of eculizumab will be given up to 48 hours post-partum, with a dose that is dependent on the dosing schedule (i.e. whether the last dose is given within the 4-week induction period or is during the maintenance phase).
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Eculizumab Intravenous Solution
  Other Names: Soliris

SUMMARY:
This is a Phase II, single arm, open-label study to determine if treatment with eculizumab prolongs pregnancy compared to historical controls in women with preeclampsia between 23-30 weeks gestation.

DETAILED DESCRIPTION:
The purpose of this study is to determine if eculizumab is an effective treatment to prolong pregnancy in women with preeclampsia, compared to a historical control group of women that received standard of care alone. Eligible subjects will be women with preeclampsia before 30 weeks gestation, who have been deemed suitable for prolongation of pregnancy.

The primary research procedure is administration of the study drug, eculizumab, by intravenous infusions weekly for four weeks, then every other week. Eculizumab is approved by the FDA for the treatment of women with atypical hemolytic uremic syndrome and paroxysmal nocturnal hemoglobinuria and is frequently used in pregnant women with these disorders. However, eculizumab is considered investigational in this study because it has not been approved by the FDA for use in patients with preeclampsia. Subject participation will last approximately 8-12 weeks on average, and the study drug will be continued until 48 hours after delivery in the treatment arm. All subjects will be followed at 2 weeks and 6 weeks after delivery to assess maternal and neonatal outcomes. A later visit may be required to complete the meningococcal vaccine schedule.

The investigators believe that eculizumab will prolong pregnancy in women with preeclampsia diagnosed before 30 weeks gestation with overactive complement. As there is no effective treatment for preeclampsia other than delivery currently, women with preeclampsia before 30 weeks gestation are managed using a "watch and wait" approach (i.e., expectant management). Due to the unpredictable nature of preeclampsia, expectant management places mother and child at significant risk until delivery occurs. Eculizumab may be an improvement over current standard of care as it provides a treatment option for patients who would otherwise be managed with expectant management alone. If the study aims are achieved, eculizumab will emerge as an effective treatment option for women with preeclampsia.

ELIGIBILITY:
Inclusion criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures & availability for study duration
3. Biologically female, aged ≥13, body weight ≥40kg
4. Diagnosed with preeclampsia between 23-29+6/7 weeks gestation, by following criteria:

   1. Blood pressure ≥160 mmHg systolic or ≥110 mmHg diastolic OR
   2. Blood pressure ≥140 mmHg systolic or ≥90 mmHg diastolic and at least one of the following

   i. Proteinuria (spot protein/creatinine ≥0.3mg/mg or 24Hr protein ≥300 mg) ii. Platelet count <100,000/μl iii. Aspartate or alanine transaminase >2x upper limit of normal iv. Creatinine >1.1 mg/dl or oliguria v. Pulmonary edema
5. Ability to take intravenous medication and be willing to adhere to the eculizumab regimen
6. Ability to receive meningococcal vaccine and be willing to adhere to antibiotic regimen

Exclusion Criteria:

An individual who meets any of the following criteria prior to enrollment will be excluded from participation in this study:

1. Known allergic reactions eculizumab or meningococcal vaccine
2. Febrile illness within prior 2 weeks
3. Treatment with another investigational drug within previous 6 months
4. Inpatient expectant management for preeclampsia >72 hours prior to enrollment
5. Fetal contraindication to expectant management of pregnancy
6. Platelet count <50,000/μl
7. Diagnosis of hemolysis, elevated liver enzymes, low platelet count (HELLP) syndrome

   * Must meet all of the following criteria to be excluded: LDH >600 U/L, platelet count < 100,000/μl, AST >2x upper limit of normal, ALT >2x upper limit of normal
8. Diagnosis of Eclampsia
9. Diagnosis of Placental abruption
10. Intrauterine fetal demise
11. Coagulopathy (INR ≥ 1.5)
12. Fibrinogen <200 mg/dl
13. Persistent, severe headache unresponsive to medications
14. Persistent, severe visual disturbances
15. Persistent, severe epigastric or RUQ pain unresponsive to medications
16. Diagnosis of Systemic lupus erythematosus
17. Diagnosis of Anti-phospholipid antibody syndrome
18. Diagnosis of Atypical hemolytic uremic syndrome
19. Diagnosis of Paroxysmal nocturnal hemoglobinuria
20. Known complement deficiency
21. Diagnosis of Venous thromboembolism active or within 6 months of enrollment
22. Diagnosis of Human immunodeficiency virus (HIV)
23. Diagnosis of Hepatitis C virus (active viremia)
24. Diagnosis of Cancer (not in remission)
25. History of Solid organ transplant
26. Systemic viral or bacterial infection (active, untreated)
27. Active use of eculizumab at time of enrollment
28. Contraindication to eculizumab treatment or complement system blockade
29. Contraindication to meningococcal vaccine
30. Body weight <40kg
31. Age <13
32. Neutropenia (<1500/mm3)
33. Gonorrhea, chlamydia, or syphilis in current pregnancy
34. Illicit substance use in current pregnancy
35. Currently homeless or incarcerated
36. Alcoholism
37. Liver cirrhosis
38. Insulin dependent diabetes
39. Active use of immunosuppressive therapies, other than use of corticosteroids for fetal lung maturity
40. Use of prophylactic or therapeutic heparin, or low molecular weight heparin, in pregnancy for hypercoagulable condition

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burwick, MD, MPH, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eculizumab
Started | 2
Completed | 1
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eculizumab
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 37.5 [35 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Latency (in Days) From Enrollment to Delivery
Description: The difference in mean number of days (latency) from enrollment in the study (or hospital admission for controls) to delivery between participant receiving eculizumab compared to historical controls.
  * For treatment-arm participants latency is determined from enrollment to delivery.
  * For historical controls latency is determined from hospital admission (or initial diagnosis for controls hospitalized for other indication) for preeclampsia until delivery.
  * Subjects and historical controls all defined as women with preeclampsia between 23-30 weeks gestation.
Time Frame: 24 months
Population: 1 enrolled subject withdrew participation before delivery. A second subject withdrew consent after delivery.
  Data supporting the primary and secondary outcomes were not collected from the two enrolled subjects. Historical controls were not identified for this terminated study, thus this Outcome Measure cannot be reported.
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Composite Adverse Maternal Outcomes
Description: The difference in the composite number of adverse maternal outcomes between subjects receiving eculizumab compared to historical controls
  •Adverse maternal outcomes directly attributed to preeclampsia defined as the following: syndrome of hemolysis, elevated liver enzyme, and low platelet count (HELLP), eclampsia, placental abruption, stroke, venous thrombosis or pulmonary embolism, pulmonary edema, posterior reversible encephalopathy syndrome, postpartum hemorrhage (>1000 cc), blood transfusion, admission to the intensive care unit, acute kidney injury, acute tubular necrosis, dialysis, or death
Time Frame: 24 months
Population: as for outcome 1
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Composite Adverse Neonatal Outcomes
Description: The difference in the composite number of adverse neonatal outcomes between subjects receiving eculizumab compared to historical controls.
  •Adverse neonatal outcomes directly attributable to preeclampsia or indirectly attributable due to preterm delivery due to preeclampsia defined as the following: Respiratory distress syndrome, bronchopulmonary dysplasia, intraventricular hemorrhage, retinopathy of prematurity, necrotizing enterocolitis, seizure, hypoxic-ischemic encephalopathy, metabolic acidosis, infection, sepsis, previously unrecognized major malformation detected at birth, patent ductus arteriosus requiring indomethacin, or death.
Time Frame: 24 months
Population: 1 enrolled subject withdrew participation before delivery. A second subject withdrew consent after delivery. 1 subject's neonate died due to extreme prematurity, which was unrelated to receiving the study drug.
  Data supporting the primary and secondary outcomes were not collected from the two enrolled subjects. Historical controls were not identified for this terminated study, thus this Outcome Measure cannot be reported.
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Changes in Blood and Urine Concentrations of Terminal Complement Protein C5a Before and After Each Treatment.
Description: The Difference in the concentration of C5a in blood and urine, before treatment ( ex. visit day 1) compared to after treatment in each participant receiving eculizumab.
  •Concentrations of C5a in blood and urine will be determined by enzyme linked immunosorbent assays (ELISA).
Time Frame: 24 months
Population: Assays for research lab samples were not done as the study was prematurely halted. Data supporting the primary and secondary outcomes were not collected from the two enrolled subjects, thus the data could not be reported.
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Changes in Blood and Urine Concentrations of Terminal Complement Protein C5b-9 Before and After Each Treatment.
Description: The difference in blood and urine concentrations of C5b-9, before treatment ( ex. visit day 1) compared to after treatment in each participant receiving eculizumab.
Time Frame: 24 months
Population: as for outcome 4
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Changes in Blood and Urine Concentrations of Complement Protein CD59 Before and After Each Treatment.
Description: The difference in blood and urine concentrations of CD59, before treatment ( ex. visit day 1) compared to after treatment in each participant receiving eculizumab.
Time Frame: 24 months
Population: as for outcome 4
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Aspartate and Alanine Transaminase Concentration Before and After Each Treatment.
Description: Differences in the concentration of aspartate and alanine transaminase (U/L) will be compared before treatment (ex. visit day 1) and after treatment in each participant receiving eculizumab.
Time Frame: 24 months
Population: as for outcome 4
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

8. Secondary Outcome: Hemoglobin Concentration Before and After Each Treatment.
Description: Differences in the concentrations of measures of hemoglobin will be compared before treatment (ex. visit day 1) and after treatment in each participant receiving eculizumab.
Time Frame: 24 months
Population: as for outcome 4
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

9. Secondary Outcome: Platelet Count Before and After Each Treatment.
Description: Differences in the platelet count will be compared before treatment (ex. visit day 1) and after treatment in each participant receiving eculizumab.
Time Frame: 24 months
Population: as for outcome 4
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

10. Secondary Outcome: Lactate Dehydrogenase Concentration Before and After Each Treatment.
Description: Differences in the concentration of serum lactate dehydrogenase will be compared before treatment (ex. visit day 1) and after treatment in each participant receiving eculizumab.
Time Frame: 24 months
Population: as for outcome 4
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

11. Secondary Outcome: Serum Creatinine Before and After Each Treatment.
Description: Differences in the concentration of serum creatinine will be compared before treatment (ex. visit day 1) and after treatment in each participant receiving eculizumab.
Time Frame: 24 months
Population: as for outcome 4
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

12. Secondary Outcome: Urine Protein Concentration Before and After Each Treatment.
Description: Differences in urine protein concentration will be compared before treatment (ex. visit day 1) and after treatment in each participant receiving eculizumab.
Time Frame: 24 months
Population: as for outcome 4
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

13. Secondary Outcome: Ratio of Urine Protein to Urine Creatinine Before and After Each Treatment.
Description: Differences in the ratio of urine protein concentration to urine creatinine concentration will be compared before treatment (ex. visit day 1) and after treatment in each participant receiving eculizumab.
Time Frame: 24 months
Population: as for outcome 4
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

14. Secondary Outcome: Serum Concentration of Soluble Fms-like Tyrosine Kinase 1 (sFlt-1) Before and After Each Treatment.
Description: Differences in the concentration of soluble fms-like tyrosine kinase 1 (sFlt-1) will be compared before treatment (ex. visit day 1) and after treatment in each participant receiving eculizumab.
Time Frame: 24 months
Population: as for outcome 4
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

15. Secondary Outcome: Serum Concentration of Placental Growth Factor (PlGF) Before and After Each Treatment.
Description: Differences in the concentration of placental growth factor (PlGF) will be compared before treatment (ex. visit day 1) and after treatment in each participant receiving eculizumab.
Time Frame: 24 months
Population: as for outcome 4
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

16. Secondary Outcome: Serum Ratio of Soluble Fms-like Tyrosine Kinase 1 (sFlt-1) Concentration to Placental Growth Factor (PlGF) Concentration (sFlt-1/PlGF) Before and After Each Treatment.
Description: Differences in the serum ratio of soluble fms-like tyrosine kinase 1 (sFlt-1) concentration to placental growth factor (PlGF) concentration (sFlt-1/PlGF) will be compared before treatment (ex. visit day 1) and after treatment in each participant receiving eculizumab.
Time Frame: 24 months
Population: as for outcome 4
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

17. Secondary Outcome: Serious Adverse Events
Description: Assessment of serious adverse events in eculizumab treatment arm compared with historical controls.
  1. Neisseria meningitidis infection or development of invasive meningococcal disease, Neisseria gonorrhoeae, Neisseria sicca/subflava, and Neisseria spp unspecified and Aspergillus infections.
  2. Graded clinical and laboratory abnormalities, according to the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS; DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1. [July 2017].
Time Frame: 24 months
Population: as for outcome 1
Arm/Group | Eculizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 months
Description: 2 subjects enrolled in the study; 1 subject withdrew before study procedures were completed
Arm/Group | Eculizumab
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=2)
Neonatal death (General disorders) | 1 (1) — Neonatal death due to prematurity

LIMITATIONS AND CAVEATS:
The PI, Dr. Richard Burwick left the institution where this research was being conducted in April 2022 and study activity halted at that time. Two subjects were consented to participate in the study and one withdrew participation before study procedures were completed. Study Funding was terminated by Sponsor.

Dr. Karumanchi is a co-investigator in this study who has been named as the Responsible Party within the PRS system solely for the purpose of reporting the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT04725812/Prot_SAP_002.pdf
  • Informed Consent Form (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT04725812/ICF_003.pdf